CLINICAL TRIAL: NCT06683118
Title: A PROSPECTIVE, MULTI-CENTER, OPEN-LABEL, SUPERIORITY, RANDOMIZED, CONTROLLED REGISTRATION TRIAL OF THE RAPAMYCIN NEUROVASCULAR BALLOON CATHETER FOR THE TREATMENT OF SYMPTOMATIC CEREBRAL ATHEROSCLEROTIC STENOSIS
Brief Title: Registration Trial of the Drug-coated Balloon for the Symptomatic Cerebral Atherosclerotic Stenosis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort NeuroTech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JUJI-2023-01-CIP-00
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Atherosclerotic Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental)
  Interventions: Device: Rapamycin neurovascular Balloon Catheter
- control group (Active Comparator)
  Interventions: Device: Conventional Balloon

INTERVENTIONS:
Device: Rapamycin neurovascular Balloon Catheter — Drug-coated balloon for the symptomatic cerebral atherosclerotic stenosis
  Arms: experimental group
Device: Conventional Balloon — Conventional Balloon for the symptomatic cerebral atherosclerotic stenosis
  Arms: control group

SUMMARY:
The purpose of the trail is to determine whether DCB is superior to conventional balloon in treating cerebral atherosclerotic stenosis

ELIGIBILITY:
Incsion Criteria:

* Age 18 to 80 years old at informed consent signing.
* Symptomatic atherosclerotic stenosis of cerebrovascular arteries with ≥70% stenosis.
* Medication ineffective.
* modified Rankin Scale(mRS) score≤2.
* The subject or guardian is able to understand the purpose of the study, is willing to participate and has given written informed consent.

Exclusion Criteria:

* History of acute ischemic stroke within 2 weeks;
* Stenosis due to non-atherosclerotic lesions such as arterial dissection, Moya-Moya disease and vasculitic disease;
* Target vessels complete occlusion or with thrombus in target vessels;
* Target vessel with severe calcification or distortion that making interventional device is difficult to place;
* History of stenting in the target artery;
* Target vessel restenosis following stenting or balloon angioplasty;
* Combined with other lesion with ≥70% stenosis in target vessel.
* Residual stenosis ≥50% or vessel dissection with obvious blood flow restriction occurs after predilation.
* Combined with intracranial tumour, arteriovenous malformation or aneurysm of the target vessel.
* History of intracranial hemorrhage within 90days.
* Presence of severe systemic diseases that cannot tolerate surgery, such as severe liver and kidney dysfunction;
* Contraindication to the use of anticoagulants and antiplatelet agents, such as sllergy to anticoagulants and antiplatelet agents, active bleeding or coagulation disorders;
* Allergic to contrast agents or rapamycin;
* Pregnant or lactating women;
* Participating or intending to participate in any other drug/device clinical trials;
* Life expectancy <1 year;
* Any other conditions that the investigator deems the patient unsuitable for enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2025-07-27 (Estimated); Study Completion 2026-07-27 (Estimated)

PRIMARY OUTCOMES:
Target lesion restenosis rate at 6 month postoperative | 180±30days
  The primary endpoint was the restenosis rate at 6 month postoperatively. Restenosis was defined as ≥50% measured stenosis of the target lesion by imaging according to WASID method.

SECONDARY OUTCOMES:
Technical succeed rate | Intraoperation
  defined as smooth delivery of the device to the target lesion and successful dilatation, unloading, and retraction
Target vascular-related stroke or death at 30 days postoperatively | 30±7days
Any stroke or death at 30 days postoperatively | 30±7days
Target vascular-related stroke or death at 6 month postoperatively | 180±30days
Any stroke or death at 6 month postoperatively | 180±30days
Target vascular-related stroke or death at 12 month postoperatively | 360±60days
Any stroke or death at 12 month postoperatively | 360±60days

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tiantan Hospital Affiliated of Peking University, Beijing, Beijing Municipality
  - Huashan Hospital Affiliated of Fudan University, Shanghai, Shanghai Municipality